CLINICAL TRIAL: NCT05439681
Title: Hs-Troponin T Kinetics in Patients Treated With MCO Membranes Compared to High-flux, Low-flux Membranes and HDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: TropT-HD
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Troponin T
Keywords: hemodialysis; low-flux dialysis; high-flux dialysis; medium cut-off membrane

STUDY DESIGN:
Intervention Model Description: Randomized controlled four-treatment, four-period crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MCO - low flux - high flux - HDF (Experimental): Patients who are on hemodialysis will be treated with four different hemodialysis sessions:
  * Treatment 1: MCO membrane
  * Treatment 2: low flux membrane
  * Treatment 3: high flux membrane
  * Treatment 4: HDF treatment with high flux membrane The order of the treatment regimens with the different membranes will be randomized.
  Interventions: Device: Theranova 400; Device: FX 10; Device: FX CorDiax 800; Device: HDF
- low flux - high flux - MCO - HDF (Experimental)
  Interventions: Device: Theranova 400; Device: FX 10; Device: FX CorDiax 800; Device: HDF
- high flux - HDF - low flux - MCO (Experimental)
  Interventions: Device: Theranova 400; Device: FX 10; Device: FX CorDiax 800; Device: HDF
- HDF - MCO - high flux - low flux (Experimental)
  Interventions: Device: Theranova 400; Device: FX 10; Device: FX CorDiax 800; Device: HDF

INTERVENTIONS:
Device: Theranova 400 — medium cut off (MCO) membrane
Device: FX 10 — low-flux membrane
Device: FX CorDiax 800 — high-flux membrane
Device: HDF — hemodiafiltration

SUMMARY:
In this study, 24 prevalent hemodialysis patients will undergo four regular hemodialysis sessions during which four different treatments will be performed.

* Treatment 1: MCO membrane (=medium cut off)
* Treatment 2: low flux membrane
* Treatment 3: high flux membrane
* Treatment 4: HDF(=hemodiafiltration) treatment with high flux membrane

So far, there is no data on cardiac bioenzyme levels during hemodialysis on the MCO membrane, thus, a acute elevation during hemodialysis might be mitigated by increased clearance.

DETAILED DESCRIPTION:
Patients who are on hemodialysis will be included in this study. After obtaining informed consent, patients will be treated with four different hemodialysis sessions:

* Treatment 1: MCO membrane (=medium cut off)
* Treatment 2: low flux membrane
* Treatment 3: high flux membrane
* Treatment 4: HDF(=hemodiafiltration) treatment with high flux membrane The order of the treatment regimens with the different membranes will be randomized in four sequences (Williams design).

Sequence 1: MCO, low flux, HDF, high flux Sequence 2: low flux, high flux, MCO, HDF Sequence 3: high flux, HDF, low flux, MCO Sequence 4: HDF, MCO, high flux, low flux Dialysis treatment will be standardized according to our clinic standard. Dialysis fluid temperature will be set to 1.0°C below the patient's body temperature, which will be assessed by auricular thermometers, to achieve maximal hemodynamic stability. Dialysis fluid composition will be standardized to calcium of 1.25mmol/L, bicarbonate of 30mmol/L, and a variable potassium and sodium concentration, depending on the patients' plasma potassium and sodium concentration.

Ultrafiltration volume will be set according to the caretaking provider.

Membranes used in the study will be FX CorDiax 10, 800 (Fresenius Medical Care, Bad Homburg vor der Höhe, Germany) and Theranova 400 (Baxter, Deerfield, Illinois, USA). We will perform the analysis only in mid-week dialysis due to the following reasons: First, hemodynamic stability is most often compromised during the first treatment of the week, due to the need of large volumes of ultrafiltration and, second, because we assume that troponin T levels reach a steady state 48 hours after the last dialysis session.

Patients undergo their routine dialysis schedule, only the membrane will be changed.

In each session, blood samples will be taken at the start of dialysis, after 1 and after 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years of age
* End stage kidney disease patient undergoing hemodialysis
* Written consent of the participant after being informed

Exclusion Criteria:

* No informed consent was obtained
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Troponin T - relative - 1 hour | 1 hour after start of hemodialysis
  Relative change from baseline (pre-treatment) to after 1 hour of hemodialysis in high sensitivity cardiac troponin T, assessed by Roche Elycsys Assay.

SECONDARY OUTCOMES:
Troponin T - relative - 4 hours | 4 hours after start of hemodialysis
  Relative change of high sensitivity cardiac troponin T from baseline to after completion of hemodialysis
Troponin I - relative - 1 hour and 4 hours | 1 hour and 4 hours after start of hemodialysis
  relative change of high sensitivity cardiac troponin I from baseline to after 1 hour and after completion of hemodialysis
Troponin T - absolute - 1 hour and 4 hours | 1 hour and 4 hours after start of hemodialysis
  absolute difference of high sensitivity cardiac troponin T from baseline to after 1 hour and after completion of hemodialysis
Troponin I - absolute - 1 hour and 4 hours | 1 hour and 4 hours after start of hemodialysis
  absolute difference of high sensitivity cardiac troponin I from baseline to after 1 hour and after completion of hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Kirsch, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No